CLINICAL TRIAL: NCT06495567
Title: Creatine Supplementation for CBS-related Homocystinuria: A Proof-of-concept Study in Healthy Adults
Brief Title: Proof of Concept Creatine Supplementation for Homocystinuria Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Rajavel Elango, PhD, Associate Professor, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H23-02515
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Homocystinuria
MeSH Terms: conditions — Homocystinuria | interventions — Creatine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline - no creatine supplementation (Experimental): Each participant will complete a baseline study day. For 7 days prior to the study day each participant will eat a controlled diet of 1g protein/kg body weight/day.
  Interventions: Dietary Supplement: Dietary methionine tracer and protein intake
- Treatment - Creatine Supplementation 20mg (Experimental): Each participant will complete a supplemented study day. For 7 days prior to the study day each participant will eat a controlled diet of 1g protein/kg body weight/day, and the provided 20mg creatine supplement.
  Interventions: Dietary Supplement: Creatine; Dietary Supplement: Dietary methionine tracer and protein intake

INTERVENTIONS:
Dietary Supplement: Creatine — For 7 days, participants will take a 20mg creatine supplement each day.
  Arms: Treatment - Creatine Supplementation 20mg
Dietary Supplement: Dietary methionine tracer and protein intake — On the study days participants will ingest 8 hourly meals of controlled amino acid intake, fortified with the necessary macronutrients. Each meal will provide one-twelfth of the participants' daily energy requirements as estimated by 1.5 x Resting Energy Expenditure (REE) and adequate protein at 1.0 g/kg/d, to maintain a metabolic steady state. The meals are in the form of a crystalline amino acid protein shake, and protein-free cookies.

SUMMARY:
Homocystinuria is a rare and inherited metabolic disorder, people with this condition don't have an enzyme needed to break down an amino acid called homocysteine. When the body can't break down the homocysteine made from another amino acid methionine, it becomes toxic to the heart, brain, and bones. We are constantly eating methionine, a building block of protein, so a common treatment is eating a low-protein diet with medical foods and vitamin pills. This can be hard to follow due to bad tastes and missing out on foods a person enjoys, especially in children.

The goal of this study is to provide participants with a supplement containing creatine, another amino acid related to methionine and homocysteine, and learn if it lowers homocysteine production in healthy adult men. We would ultimately like to see if creatine supplements are a potential alternate treatment of Homocystinuria in this proof of concept study, before studying individuals with the condition.

Researchers in this study want to know:

* How does the bodies digestion of isotope methionine change in breath and urine when creatine is taken in healthy young adult men?
* How do levels of homocysteine, methionine and related metabolites change in the blood when creatine is taken by healthy young adult men?

Participants will:

* Complete two (2), 8-hour study days on-site.
* Eat a lower protein diet for one (1) week before the first study day, and eat a lower protein diet with creatine supplements for one (1) week before the second study day.
* During both study days eat special hourly meals of controlled amino acids and nutrients, along with a methionine isotope. (An isotope is a stable labelled amino acid that is colourless, odorless, tasteless, and safe for consumption. In the lab we can detect this isotope in breath and urine samples collected during the study day).
* Provide samples of breath, urine and blood. (Researchers will also take body measurements (height weight), and use non-invasive tests to measure body composition and energy needs).

DETAILED DESCRIPTION:
Homocystinuria is a rare but potentially serious inherited condition due to cystathionine beta-synthase (CBS) deficiency which causes accumulation of homocysteine and its precursor methionine.

Our hypothesis is that high doses of orally supplemented creatine will lead to a reduction of endogenous production of homocysteine. Our hypothesis is based on the tight association of the metabolic pathways for creatine synthesis and the synthesis of S-adenosylhomocysteine (SAH) which is the immediate precursor of homocysteine. Suppression of endogenous creatine synthesis through provision of exogenous creatine will lead to reduced production of SAH and thus homocysteine.

Our objectives are:

1. To test endogenous methionine turn over using stable isotope technique in response to creatine supplementation in healthy young adult men
2. To test changes in blood levels of homocysteine, S-adenosylmethionine (SAM), SAH and methionine as well as creatine metabolites dependent on creatine supplementation

To test the endogenous methionine turn over in response to creatine supplementation we will use stable isotope techniques utilizing labelled carbon (13C), as 1-13C-Methionine. The tracer will be given along with protein shakes composed of specific amounts of protein (1g/kg/d) and its metabolic fate can be tracked by measuring 13C labelled carbon dioxide (CO2) in breath samples and 13C species in urine with mass spectrometer. Stable isotopes have been used previously and are currently being used for metabolic studies in healthy children and adults, including pregnancy. Our Lab has special experience with this technique and has used it for the study of other inborn errors of metabolism. For the measurement of plasma levels of homocysteine, methionine, SAM, SAH, creatine and its intermediates we will use mass spectrometry, employing well established methods in our lab.

We will perform a baseline study (without previous creatine supplementation and a treatment study (with previous creatine supplementation) in two separate study days. Participants will take a diet providing 1 gram of protein /kg/day for 7 days prior to the respective study. For the treatment, study participants will additionally take 20 grams of creatine per day for 7 days. On the study days probands will take hourly experimental meals containing the tracer methionine and breath samples and urine samples will be collected to determine 13C species coming from the ingested methionine. We will collect blood during the 6th hour of the study to determine methionine and creatine related metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Cis-male
* Men who are classified as normal body weight and BMI (18.5-25kg/m2)
* Free of any concurrent illness (cold, flu, vomiting etc.)
* Not be claustrophobic (we will place a clear hood, which can easily be removed, over your head for approximately 20 min to measure your energy expenditure)
* Not be enrolled in any other research studies (as this may affect our study results)

Exclusion Criteria:

* Men not in good health or have a metabolic, neurological, genetic, or immune disorder, including diabetes, hypoglycemia, hypertension and current or past history of kidney disease
* Men who have food allergies/sensitivities/intolerances to egg, corn, diary etc.
* Men who have current or recent past history of ingesting creatine supplements
* Men who are smokers
* Men who are following a non-traditional dietary pattern (e.g. Keto diet, Atkins diet, paleo diet, intermittent fasting, strict vegan, calorie restricted diet etc.)

Ages: 19 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Carbon 13 Oxidation | 8 hours
  Urine and breath samples will be collected to measure the rate of L-[1-13C]methionine oxidation

CONTACTS AND LOCATIONS:
Overall Officials: Rajavel Elango, PhD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital Research Institute, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided